CLINICAL TRIAL: NCT02968134
Title: Single Dose Population Pharmacokinetics of Intravenous Posaconazole in Critically Ill Patients
Acronym: POSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Brisbane and Women's Hospital (Other Government)
Collaborators: The University of Queensland (Other)
Responsible Party: Principal Investigator, Jason Roberts, Professor, Royal Brisbane and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HREC/16/QRBW/377
Record Dates: First submitted 2016-11-15; First posted 2016-11-18 (Estimated); Results first posted 2018-07-09 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Systemic Fungal Infections
MeSH Terms: interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posaconazole (Other): The study will enrol eight patients with presumed or confirmed systemic fungal infections, who are admitted to ICU
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — A single dose of 300mg intravenous posaconazole will be administered and blood samples will be taken prior to start of infusion, at 15,45,75minutes, 3,5,8,12,18,24,30,36 and 48 hours.
  Other Names: Noxafil

SUMMARY:
The purpose of this study is to try to find out how critically ill patients receiving the anti fungal medication, posaconazole, process it in their body. Investigators would like to study if the recommended doses of posaconazole achieve adequate concentrations in the patients blood to treat fungal infections.The disease process in critically ill patients can profoundly influence the concentration of anti fungal medication in the blood. The process by which a drug travels through the body in blood, how it is broken down and removed by the body is called pharmacokinetics (PK).

This information is important to know because if antifungal levels are low in the blood, the fungal infection has an opportunity to become resistant to the antifungal medication which can lead to the medication being less effective against the fungal infection potentially exposing future patients with infection to a limited range of effective antifungals.

Investigators can measure the PK by taking blood samples at specific times after the anti fungal medication is given.

This study will enroll 8 patients who are admitted to the intensive care unit and are being treated with an antifungal medication for a fungal infection. Patients will be consented and given a single dose of posaconazole and serial blood samples will be collected just prior to the dose and at 15, 45,75 minutes during the infusion and at 3, 5, 8, 12, 18, 24, 30 36 and 48 hours . Information about the patients stay in the ICU will also be collected including blood pressure, temperature, blood test results.

DETAILED DESCRIPTION:
Posaconazole is a new extended spectrum triazole active against a range of yeasts and molds including Aspergillus, Candida, Coccidioides, Cryptococcus neoformans, Fusarium, and Zygomycetes. It may be used for the prevention of invasive fungal infections in immunocompromised patients including febrile neutropenic patients and those receiving immunosuppressant drugs for graft-vs-host disease during stem cell transplantation. It may also be used for treatment of systemic fungal infections.The use of posaconazole in ICU patients has been limited to stable patients to ensure reliable bioavailability from the oral formulations. Oral formulations have important limitation in that they cannot be used in critically ill patients who may be unable to take oral doses or bioavailability may be compromised due to erratic absorption. Recently, an intravenous (IV) formulation has been developed to address these limitations. Initial pharmacokinetic (PK) investigations of the IV formulation were conducted in hematology patients, with further data in other patient populations still forthcoming; particularly in the critically ill where the IV formulation would probably be used most frequently.

Most of the available PK data for posaconazole is from non-critically ill patients who received the oral formulation. Although the absorption phase of the kinetics is not relevant for the IV formulation, data on the distribution, metabolism and elimination properties would still be informative of the IV kinetics. The tissue distribution of posaconazole is extensive with a very large volume of distribution owing to its high lipophilicity. It is highly bound to plasma proteins (98-99%) and therefore very likely to be affected by the variable changes in plasma protein concentration in critically ill patients. The major elimination pathway of posaconazoleis through biliary excretion (about 77%) of mainly the unchanged parent compound and the rest through renal execration of as a glucuronide conjugate.

A number of studies have described PK variability of posaconazole due to altered absorption/bioavailability which can frequently result in sub-therapeutic plasma concentrations, forming strong case for therapeutic drug monitoring. Nonetheless, it is unclear whether the observed low concentrations can also be explained, at least in part, by other factors such as disease-related PK changes or if the obvious plausibility of altered absorption has masked such investigations. Most population PK models described so far are based on one compartment models, which do not reveal if the observed variability in concentrations is due to changes in PK parameters such as volume of distribution or clearances. The influence of disease state on these PK parameters has been extensively described for several antimicrobials in the critically ill patient populations. Although data on the new IV formulation of posaconazole in this patient population is lacking, there is evidence from previous PK studies on the oral formulation that PK variability not observed in healthy study participants was observed in patients with invasive fungal infections, although it was explained primarily in relation to altered bioavailability from the oral formulation. In surgical ICU patients low plasma concentration of posaconazole were observed, after administration via nasogastric tube. Similar findings were reported in general ICU patients. Although the explanation in these reports was again the irregular absorption, the influence of other pathologic changes remains to be investigated. A PK evaluation of IV posaconazole in critically ill patients, not confounded by the absorption factor, would reveal if there is any pathophysiology-induced PK alteration. Such a study will also give insight into the dose-exposure relationships and optimal treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Admission for ICU care
* The presence of suspected or confirmed fungal infection requiring systemic antifungal therapy
* Presence of central venous access for drug administration

Exclusion Criteria:

* Age < 18 years
* Pregnancy
* Prescription of drugs that are known to interact with posaconazole
* Oral posaconazole use within the last two week prior to enrolment
* Documented history of drug reaction to the triazole antifungal medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-05-21 (Actual); Study Completion 2017-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Roberts, BPharm, Principal Investigator — Royal Brisbane and Womens Hospital

IPD SHARING:
Plan to Share IPD: No
De-identified data for all primary and secondary endpoints will be reported as a collective data set. Individual results will not be reported.

REFERENCES:
- [Result] Sime FB, Stuart J, Butler J, Starr T, Wallis SC, Pandey S, Lipman J, Roberts JA. Pharmacokinetics of Intravenous Posaconazole in Critically Ill Patients. Antimicrob Agents Chemother. 2018 May 25;62(6):e00242-18. doi: 10.1128/AAC.00242-18. Print 2018 Jun. PMID 29581122

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posaconazole
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Posaconazole
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Body mass index calculated in kg/m2
  kg/m^2 | 22.6 [20.2 to 29.7]
Acute Physiology and Chronic Health Evaluation II Score [Median (Inter-Quartile Range); unit: units on a scale] — Acute Physiology and Chronic Health Evaluation II [APACHE II] score on ICU admission was calculated from 12 routine physiologic measurements using standard approach. APACHE II score ranges from 1 to 71, with higher scores correlating with increased risk of mortality. For a detailed description, please refer to Crit Care Med. 1985 Oct;13(10):818-29.
  units on a scale | 17 [17 to 24]
Serum creatinine [Median (Inter-Quartile Range); unit: umol/L] | 106 [78 to 179]
Urinary creatinine clearance [Median (Inter-Quartile Range); unit: mL/min] | 74 [53 to 109]
Serum albumin [Median (Inter-Quartile Range); unit: g/L] | 20 [18 to 20]
ALT [Median (Inter-Quartile Range); unit: IU/mL] — Alanine transaminase
  IU/mL | 53 [28 to 60]
AST [Median (Inter-Quartile Range); unit: IU/mL] — Aspartate transaminase
  IU/mL | 47 [38 to 130]
ALP [Median (Inter-Quartile Range); unit: IU/mL] — Alkaline phosphatase
  IU/mL | 75 [63 to 108]
Total bilirubin [Median (Inter-Quartile Range); unit: umol/L] | 11 [10 to 20]
INR [Median (Inter-Quartile Range); unit: ratio] — International normalized ratio
  ratio | 1.3 [1.3 to 1.4]

OUTCOME MEASURES:

1. Primary Outcome: Posaconazole Exposure Described as Area Under the Total Plasma Concentration-time Curve From Time Zero to Infinity After a Single Dose
Description: The primary outcome is plasma posaconazole exposure expressed as the area under the total plasma concentration-time curve from time zero to infinity resulting from a single dose of 300 mg of posaconazole administered intravenously.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 8
ng*h/mL | 17932 [13823 to 27905]

2. Primary Outcome: Posaconazole Exposure Expressed as Area Under the Unbound Concentrations-time Curve From Time Zero to Infinity
Description: This is a measure of free posaconazole ( not bound to plasma proteins) exposure in the plasma. This is an important measure of exposure because its the free concentration that distributes into targets sites of infection to produce clinical effect.
Time Frame: 48 hours
Measure: Median (Inter-Quartile Range); unit: ng*h/mL
Arm/Group | Posaconazole
Number analyzed (Participants) | 8
ng*h/mL | 97.2 [72.8 to 134.8]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over one and half year of patient enrolment.
Arm/Group | Posaconazole
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=8)
Death (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT02968134/Prot_SAP_000.pdf